CLINICAL TRIAL: NCT03034005
Title: The RECONSTRUCT Study - Reconstructing Disease Mechanisms in Asthma
Acronym: RECONSTRUCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Celeste Porsbjerg, Associate Professor, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-003509-33
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids; Airway hyper-responsiveness; Airway smooth muscle; sodium-potassium pump
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with asthma (Experimental): 6 weeks treatment with 1600 ug budesonide
  Interventions: Drug: Budesonide
- Healthy Controls (No Intervention): Healthy controls to establish baseline level of Na/K pumps.

INTERVENTIONS:
Drug: Budesonide — 1600 ug inhaled daily for 6 weeks
  Other Names: Pulmicort
  Arms: Patients with asthma

SUMMARY:
This study aims to assess the effect of inhaled corticosteroids (ICS) on airway smooth muscle (ASM) Na+, K+ pumps in patients with asthma.We wish to investigate differences in Na+, K+ pump content in healthy versus asthmatic patients, whether a reduction in airway hyper-responsiveness observed in asthmatic patients treated with ICS is attributable to an increase in Na+, K+ pump content in ASM cells and compare this in patients with non-eosinophilic asthma versus eosinophilic asthma.

DETAILED DESCRIPTION:
Purpose and background

Inhaled corticosteroids and asthma phenotypes Inhaled corticosteroid (ICS) is a cornerstone in the treatment of asthma. ICS acts locally in the airways through several pathways to limit inflammation, primarily through reduction of eosinophilic inflammation.

In clinical practice however a substantial part of adult patients with asthma have no eosinophilic inflammation in the airways despite reduced lung function and increased contractility of the smooth muscles in the airways i.e., airway hyperresponsiveness(AHR). This group of patients with non-eosinophilic asthma (NEA) represents up to 50 % of adult asthmatics with even higher occurrence among patients referred to a specialist.

The effect of ICS in NEA is debated but despite lack of eosinophilic inflammation, ICS has been shown to significantly reduce AHR in patients with NEA, suggesting mechanistic pathways different from reduction in eosinophilic inflammation.

Airway smooth muscle and inhaled corticosteroids Airway smooth muscle (ASM) is the most abundant tissue type in the airways. It plays a crucial part in the pathogenesis of asthma and serves as an important target for therapy especially with β-adrenergic agents and to some extent anti-muscarinic agents, counteracting bronchoconstriction. However also ICS has been proposed to have direct action on ASM cells affecting contractility through reduction of intracellular Ca2+ or down regulation of membrane bound receptors as well as through limiting cellular proliferation and secretory function. The bronchodilating effect of β-adrenergic agents has in animal models shown to be potentiated by administration of corticosteroids.

Inhaled corticosteroids and the Na+, K+ pump Both ICS and systemically administered prednisone has been shown to increase Na+, K+ pump activity in leucocytes from patients with asthma and in both rats and humans systemically administered corticosteroid increases the amount of Na+, K+ pumps in striated muscle by 20-40 % and 30-60 % respectively. We have recently demonstrated a similar effect with ICS where a therapeutically relevant daily dose of 1600 μg budesonide, administered in the respiratory tract by inhalation, increased the amount of Na+, K+ pumps in striated muscle by 17 %.

1.1.4 The Na+, K+ pump and airway smooth muscle The Na+, K+ pump creates an inward Na+ current by removing Na+ from the intracellular lumen of cells. This may drive extrusion of Ca2+ from the lumen of the ASM cells through the Na+, Ca2+ exchanger lowering intracellular Ca2+ concentration. Since Ca2+ plays a central role in smooth muscle contraction, lower intracellular concentrations may protect against bronchoconstriction as well as the contrary might reinforce AHR.

In vitro studies have demonstrated disturbances in leucocyte Na+, K+ pump activity and increased intracellular Na+ in patients with hyperreactivity and asthma. Likewise in vitro studies of human bronchial muscle have shown increased AHR and concentrations of intracellular Ca2+ as well as decreased β-adrenergic induced relaxation of human bronchial muscle when Na+, K+ pumps are blocked.

Bronchoconstriction and airway remodeling are universal features of asthma and especially bronchoconstriction can to some extent be related to proposed disturbances in Na+, K+ pump activity and positive effects of ICS besides being anti-inflammatory is therefore suspected to be beneficial independent of cellular patterns. However the non-inflammatory effect might be more evident in patients with NEA since it is not blurred by the anti-inflammatory effect seen in patients with EA.

No studies have assessed the effect of ICS on ASM Na+, K+ pumps in patients with asthma. In the present study the investigators wish to study differences in Na+, K+ pump content in healthy versus asthmatic patients, whether a reduction in AHR observed in asthmatic patients treated with ICS is attributable to an increase in Na+, K+ pump content in ASM cells and compare this in patients with NEA versus EA.

This results in a study in two parts:

I. A comparison of the level of Na+, K+ pumps in ASM in patients with asthma vs healthy subjects.

II. A description of the association between changes in Na+, K+ pump content in ASM and change in AHR after ICS in patients with asthma.

Hypothesis Study part I: The amount of ASM Na+, K+ pumps are lower in adult patients with asthma compared to healthy subjects.

Study part II: The reduction in airway hyperresponsiveness in adult patients with asthma after treatment with ICS is related to an increase in the content of Na+, K+ pumps in ASM.

We further hypothesize that the association between the increase in Na+, K+ pumps in ASM and the change in AHR after ICS treatment is strongest in NEA versus EA.

Aim Study part I: To describe differences in ASM content of Na+, K+ pumps among healthy subjects and patients with NEA or EA respectively.

Study part II: To describe the correlation between increase in ASM content of Na+, K+ pumps and reduction in airway hyperresponsiveness to mannitol after six weeks of daily inhalation of glucocorticoid, in patients with asthma.

Perspectives Asthma is common and may be difficult to treat, especially the non-eosinophilic phenotype. This study aims to increase our understanding of pathogenic mechanisms in asthma, unrelated to inflammatory pathways. This may lead towards a shift from the current paradigm of asthma as a purely inflammatory condition, creating novel understanding of the role of ion transport regulation in the pathogenesis and treatment of asthma, ultimately revealing targets for novel treatments.

ELIGIBILITY:
Inclusion Criteria:

* Asthma as defined by GINA (www.ginasthma.org) Eosinophilic asthma: Fractional exhaled nitric oxide (FeNO) > 25 ppb (marker of eosinophilic airway inflammation) Non-eosinophilic asthma: Fractional exhaled nitric oxide (FeNO) < 25 ppb
* An FEV1 value of ≥70% of expected
* Airway hyperresponsiveness to mannitol (PD15 ≤ 315 mg)
* Not treated with oral or inhaled steroids (past 3 months)

Exclusion Criteria:

* Smoking (current smokers or a maximum of 10 pack years)
* Competing respiratory diseases
* Lower respiratory tract infection within the past 4 weeks
* Medical history with significant comorbidity (ASA>2)
* Pregnant or breastfeeding
* Hypersensitivity to study medication including Spirocort, Osmohale, Midazolam or Fentanyl
* Uncontrolled hypertension
* Acute myocardial infarction within past 6 months
* Aorta- or cerebral aneurism
* Recent abdominal operation
* Failure to comply with study protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in airway hyperresponsiveness (mannitol challenge) per change in Na+, K+ pumps content in airway smooth muscle. | 6 weeks
  Change in PD15 per chhange in NA/K ATP'ase content

SECONDARY OUTCOMES:
Change in Na+, K+ pump content in airway smooth muscle and in skeletal muscle (ρmol ouabain per g wet weight) in NEA vs. EA. | 6 weeks
  Change in Na+, K+ pump content in airway smooth muscle and in skeletal muscle (ρmol ouabain per g wet weight) in NEA vs. EA.
Change in airway hyperresponsiveness (PD15 to mannitol) in NEA vs. EA | 6 weeks
  Change in airway hyperresponsiveness (PD15 to mannitol) in NEA vs. EA

OTHER OUTCOMES:
Change in asthma control score vs in Na+, K+ pumps content in airway smooth muscle. | 6 weeks
  Change in asthma control score vs in Na+, K+ pumps content in airway smooth muscle.
Change in lung function (FEV1) vs in Na+, K+ pumps content in airway smooth muscle | 6 weeks
  Change in lung function (FEV1) vs in Na+, K+ pumps content in airway smooth muscle
Change in asthma control score in NEA vs. EA | 6 weeks
  Change in asthma control score in NEA vs. EA
Change in lung function (FEV1) in NEA vs. EA | 6 weeks
  Change in lung function (FEV1) in NEA vs. EA

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Porsbjerg, Principal Investigator — Assistant Professor
Locations (1):
- Lungemedicinsk forskningsenhed, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No